CLINICAL TRIAL: NCT04945616
Title: Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR2285 Tablets Combined With Aspirin, Clopidogrel or Ticagrelor in Healthy Subjects
Brief Title: To Evaluate the Safety and Tolerability of Combined Administration of SHR2285 Tablets With Aspirin, Clopidogrel or Ticagrelor in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SHR2285-106
Record Dates: First submitted 2021-06-01; First posted 2021-06-30 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A： Aspirin + Clopidogrel + placebo or SHR2285 (dose 1) (Experimental)
  Interventions: Drug: Aspirin、clopidogrel、placebo or SHR2285
- group B ：Aspirin + Clopidogrel + placebo or SHR2285 (dose 2) (Experimental)
  Interventions: Drug: Aspirin、clopidogrel、placebo or SHR2285
- group C： Aspirin + Ticagrelor + placebo or SHR2285 (Experimental)
  Interventions: Drug: Aspirin、ticagrelor、placebo or SHR2285

INTERVENTIONS:
Drug: Aspirin、clopidogrel、placebo or SHR2285 — groupA： Aspirin + clopidogrel + placebo or SHR2285 (dose 1) ；
  Arms: group A： Aspirin + Clopidogrel + placebo or SHR2285 (dose 1)
Drug: Aspirin、clopidogrel、placebo or SHR2285 — groupB： Aspirin + clopidogrel + placebo or SHR2285 (dose 2)
  Arms: group B ：Aspirin + Clopidogrel + placebo or SHR2285 (dose 2)
Drug: Aspirin、ticagrelor、placebo or SHR2285 — groupC： Aspirin + ticagrelor + placebo or SHR2285
  Arms: group C： Aspirin + Ticagrelor + placebo or SHR2285

SUMMARY:
The study is a single-center，randomized, doubled-blinded, placebo-controlled, Only for SHR2285 Phase I trial. This study intends to enroll 52 healthy subjects, regardless of gender. The subjects are divided into three groups: A, B, and C, with 16 cases in each of groups A and B, and 20 cases in group C.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, aged 18-55 (including boundary);
2. Body mass index (BMI) between 19 to 28 kg/m2 (including boundary), male body weight ≥50 kg and <90 kg , female body weight ≥45kg and <90kg;
3. Participant with no clinically significant findings in vital signs, physical examination, 12-lead ECG ,X-ray and laboratory parameters，etc.
4. Understand the study procedures and methods, voluntary to participate in the study and signed the informed consent.

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin/direct bilirubin > 1.2 fold ULN during screening/baseline.
2. Serum creatinine> ULN during screening/baseline.
3. Positive faecal occult blood
4. Abnormal coagulation function.
5. A clinical history of coagulation dysfunction; subjects with adverse reaction of antiplatelet drugs or anticoagulant drugs.
6. Subjects with severe head trauma or head surgery within 2 years or surgery within 3 months prior to the screening.
7. Blood donation or blood loss within 1 month≥200 mLor≥400 mL within 3 months before administration.
8. Human immunodeficiency virus antibody, syphilis serological examination, hepatitis b virus surface antigen, hepatitis c virus antibody were positive.
9. 3 months prior to screening involved in any drug or medical device clinical studies. .
10. Female subjects who did not receive contraception at least 30 days before administration and etc.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and severity of adverse events. | from the first dose to 48hours after the last dose

SECONDARY OUTCOMES:
Cmax | from Day1 to Day8 after the first dose
  Maximum observed serum concentration (Cmax) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite steady state after multiple administrations.
Tmax | from Day1 to Day8 after the first dose
  Time to maximum observed serum concentration (Tmax) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite at steady state after multiple administrations.
T1/2 | from Day1 to Day8 after the first dose
  Time to elimination half-life (T1/2) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite at steady state after multiple administrations.
AUC0-last | from Day1 to Day8 after the first dose
  Area under the plasma concentration versus time curve (AUC0-last) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite at steady state after multiple administrations.
Cmax，ss | from Day1 to Day8 after the first dose
  Steady-state peak concentration (Cmax，ss) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite at steady state after multiple administrations.
Ctrough，ss | from Day1 to Day8 after the first dose
  Steady state valley concentration (Ctrough，ss) for acetylsalicylic acid and its active metabolite salicylic acid, clopidogrel, ticagrelor and its active metabolite AR-C124910XX, SHR2285 and its active metabolite at steady state after multiple administrations.
FXI activity | from Day1 to Day8 after the first dose
  Clotting factor XI (FXI) activity
APTT | from Day1 to Day8 after the first dose
  Change of activated partial thromboplastin time (APTT) from baseline
PT | from Day1 to Day8 after the first dose
  Change of prothrombin time (PT) from baseline
INR | from Day1 to Day8 after the first dose
  Change of international normalization ratio (INR) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided